CLINICAL TRIAL: NCT05025579
Title: What is the Effect of Aerobic Exercise on Depression in Geriatric Individuals Diagnosed With Depression?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03/15/2019-74
Record Dates: First submitted 2021-08-24; First posted 2021-08-27 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Aerobic Exercise; Depression; Geriatric; Chronic Illness
Keywords: Aerobic Exercise; Depression; Geriatric; Chronic Illness
MeSH Terms: conditions — Depression; Chronic Disease | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The study, 65-75 years of age a in range, geriatric depression diagnosed with and willing to participate in the study is when individuals were included in the study. Geriatrics psychiatric disorders other than depression who, for any reason unable to ride a bike, that static man, to exercise contraindications u found my show compliance with the exercise program and to the individuals who were excluded from the study .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise group (Experimental): Considering the protocol suggested in the literature and by examining exercise samples for geriatric individuals, an exercise protocol was created. The first week started with aerobic exercises with a total of 120 minutes, and the next week increased to 160 minutes . A 6-week exercise program was planned and applied 4 days a week in which the intensity was increased gradually. People 's heart rate, blood pressure and respiratory frequency exercise program implementation before and after was recorded in the evaluation form.
  Interventions: Other: Aerobic Exercise

INTERVENTIONS:
Other: Aerobic Exercise — Since up in 2 min 10 repetitions active joint movement (while seated knee flexion and extension the ankle plantar and dorsal flexion , standing the hip flexion , extension the , abduction and adduction ) , treadmill for 3 minutes, 0.5 m / sec speed walk with and to adapt both warming bike 5 minutes, RPE ( Rating of Perceived exertion discoverable by exertion rate) will be 2/10 in a way was built.
  As aerobic exercise, the first week will be RPE 4/10 for 10 minutes, the second week with RPE 4/10 12 minutes, the third week with RPE 4/10 14 minutes, the fourth week with RPE 4/10, 16 minutes, the fifth week with RPE 5/ 2 0 will be as 18 minutes sixth week RPA 10.6 will form was done 20 minutes of exercise .
  Cooling period in the RPE 2.10 will be the 5 minute turning cycling, 5 min active range of motion exercises and stretching was done.

SUMMARY:
This study was planned to examine the effect of aerobic exercises on depression in geriatric individuals with a diagnosis of depression.

DETAILED DESCRIPTION:
In this study 67 ± 5 years of age averaged and by the physician in geriatric depression diagnosis was placed 38 sedentary geriatric subjects were included. Meet the inclusion criteria geriatric individuals information, vital signs (pulse,"beats /min", blood pressure, " mmHg ", respiration number, respiratory rate,) was recorded. Depression levels, Depression Outcome Scale- KOFDSS to and quality of life is Quality of Life Survey -EUROHIS WHO-QOL) were evaluated. 6-week, 4 days a week aerobic exercise program was applied to geriatric individuals. As aerobic exercise which included the heating and cooling cycle was started the first week and 120 minutes, 160 minutes weekend out and gradually the intensity was given as an exercise program to be increasing. Individuals from the 6-week program were re-evaluated.

ELIGIBILITY:
Inclusion Criteria:

* 65-75 years of age a in range, geriatric depression diagnosed with and willing to participate in the study is when individuals were included in the study.

Exclusion Criteria:

* Having geriatric psychiatric disorders other than depression, not being able to ride a bike for any reason, have contraindications for exercise, inability to adapt to exercise, not volunteering to participate

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
geriatric depression | before and after treatment (24 sessions, beginning and 6th. weeks)
  Change from Clinically useful depression outcome scale score at beginning and 6th. weeks

SECONDARY OUTCOMES:
Life Quality | before and after treatment (24 sessions, beginning and 6th. weeks)
  Change from World Health Organization Quality of Life Questionnaire (EUROHIS-QOL) score at beginning and 6th. weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rabia Tugba Kilic, Principal Investigator — Ankara Yildirim Beyazit University,Faculty of Health Sciences, Physiotherapy and Rehabilitation Department ANKARA, Turkey, 06760; Bonny Wamukoya Wasıke, Study Director — Ankara Yildirim Beyazit University, Faculty of Health Sciences, Physiotherapy and Rehabilitation Department; Necmiye Un Yildirim, Study Chair — Ankara Health Sciences University Department of Physical Therapy and Rehabilitation
Locations (1):
- Ankara Yildirim Beyazit University,Faculty of Health Sciences, Physiotherapy and Rehabilitation Department, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Blumenthal JA, Babyak MA, Moore KA, Craighead WE, Herman S, Khatri P, Waugh R, Napolitano MA, Forman LM, Appelbaum M, Doraiswamy PM, Krishnan KR. Effects of exercise training on older patients with major depression. Arch Intern Med. 1999 Oct 25;159(19):2349-56. doi: 10.1001/archinte.159.19.2349. PMID 10547175
- [Background] Rinaldi P, Mecocci P, Benedetti C, Ercolani S, Bregnocchi M, Menculini G, Catani M, Senin U, Cherubini A. Validation of the five-item geriatric depression scale in elderly subjects in three different settings. J Am Geriatr Soc. 2003 May;51(5):694-8. doi: 10.1034/j.1600-0579.2003.00216.x. PMID 12752847
- [Background] Egede LE, Nietert PJ, Zheng D. Depression and all-cause and coronary heart disease mortality among adults with and without diabetes. Diabetes Care. 2005 Jun;28(6):1339-45. doi: 10.2337/diacare.28.6.1339. PMID 15920049
- [Background] Lieberwirth C, Wang Z. The social environment and neurogenesis in the adult Mammalian brain. Front Hum Neurosci. 2012 May 8;6:118. doi: 10.3389/fnhum.2012.00118. eCollection 2012. PMID 22586385
- [Background] Babyak M, Blumenthal JA, Herman S, Khatri P, Doraiswamy M, Moore K, Craighead WE, Baldewicz TT, Krishnan KR. Exercise treatment for major depression: maintenance of therapeutic benefit at 10 months. Psychosom Med. 2000 Sep-Oct;62(5):633-8. doi: 10.1097/00006842-200009000-00006. PMID 11020092
- [Background] Christmas C, Andersen RA. Exercise and older patients: guidelines for the clinician. J Am Geriatr Soc. 2000 Mar;48(3):318-24. doi: 10.1111/j.1532-5415.2000.tb02654.x. PMID 10733061